CLINICAL TRIAL: NCT03794986
Title: Peer Online Motivational Interviewing for Sexual and Gender Minority Male Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000024842; AD-2018C1-11098 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-12-12; First posted 2019-01-07 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: Sexual Abuse
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: randomized comparative
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational Interviewing (Experimental): Sexual and gender minority males who are sexual abuse survivors.
  Interventions: Behavioral: Motivational Interviewing
- MI with trauma-informed SGM affirmative care (Active Comparator): MI w/trauma-informed SGM affirmative care
  Interventions: Behavioral: Trauma-informed SGM affirmative care

INTERVENTIONS:
Behavioral: Trauma-informed SGM affirmative care — All SGM male survivors who meet inclusion criteria, including significant emotional distress, will complete pre-test measures and be randomized to 6-week Motivational Interviewing (MI) delivered by peers in online groups or 6-week MI with trauma-informed, SGM affirmative care delivered by peers in online groups.
  Participants will complete pre-intervention (baseline), end of the 6-week intervention, 60- and 120-days follow-up assessments via an online survey platform, to determine if there was an increase in formal treatment engagement, and any significant changes in mental health symptomology (i.e., PTSD, depression, high-risk drinking, and illicit substance use).
  Arms: MI with trauma-informed SGM affirmative care
Behavioral: Motivational Interviewing — Major principles and tenets of Motivational Interviewing (MI) group include: Non-confrontational nature of group; environment is one of respect, safety, and encouragement of all group members; purpose is to learn about members' personal thoughts and choices and not to push an "agenda"
  Arms: Motivational Interviewing

SUMMARY:
The study will conduct a randomized comparative effectiveness trial of peer-facilitated, online, 6-week group Motivational Interviewing (MI) vs. Motivational Interviewing (MI) with a trauma-informed Sexual and Gender Minority (SGM) affirmative care approach.

DETAILED DESCRIPTION:
Through workshops and ongoing supervision/consultation, researchers will train MaleSurvivor peer leaders to competently deliver both versions of MI and conduct a randomized controlled trial comparing the two versions of MI to enhance treatment engagement in SGM male survivors with mental health problems. All SGM male survivors who meet inclusion criteria, including significant emotional distress, will complete pre-test measures and be randomized to 6-week MI delivered by peers in online groups or 6-week MI with trauma-informed, SGM affirmative care delivered by peers in online groups. Randomization will be counterbalanced by treatment status: treatment naive versus treatment-experienced (prior treatment but not within the past 60 days).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking; men who have sex with men or individuals identifying as SGM males
* Individuals who report a history of sexual abuse and individuals who self-report a minimum cut-off score of 3.0 or higher on emotional distress, using a 4-question symptom inventory.

Exclusion Criteria:

* Individuals who endorse active psychosis
* Individuals who have a cognitive dysfunction
* SGM men who report that they are currently in formal mental health counseling

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Men who have sex with men or individuals identifying as sexual gender minority (SGM) males who report a history of sexual abuse.
Enrollment: 356 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan Cook, Phd, Principal Investigator — Yale School of Medicine Department of Psychiatry
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Mandavia AD, Banducci AN, Simpson TL, Marx BP, Hawn SE, Hyde J, Ameral VE, Sistad Hall RE, Roth CE, Sarpong AA, Davenport M, Meng F, Stein MD, Livingston NA. Sex Differences in Suicide, Lethal Means, and Years of Potential Life Lost Among Veterans With Substance Use Disorder. Womens Health Issues. 2025 May-Jun;35(3):196-204. doi: 10.1016/j.whi.2025.02.002. Epub 2025 Mar 19. PMID 40113455
- [Derived] O'Doherty L, Whelan M, Carter GJ, Brown K, Tarzia L, Hegarty K, Feder G, Brown SJ. Psychosocial interventions for survivors of rape and sexual assault experienced during adulthood. Cochrane Database Syst Rev. 2023 Oct 5;10(10):CD013456. doi: 10.1002/14651858.CD013456.pub2. PMID 37795783

RESULTS

PARTICIPANT FLOW:
Groups:
- MI With Trauma-informed SGM Affirmative Care: MI w/trauma-informed SGM affirmative care
  Trauma-informed SGM affirmative care: All SGM male survivors who meet inclusion criteria, including significant emotional distress, will complete pre-test measures and be randomized to 6-week Motivational Interviewing (MI) delivered by peers in online groups or 6-week MI with trauma-informed, SGM affirmative care delivered by peers in online groups.
  Participants will complete pre-intervention (baseline), end of the 6-week intervention, 60- and 120-days follow-up assessments via an online survey platform, to determine if there was an increase in formal treatment engagement, and any significant changes in mental health symptomology (i.e., PTSD, depression, high-risk drinking, and illicit substance use).
Period: Overall Study
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Started | 178 (Randomized) | 178 (Randomized)
Partial Completion | 35 (Attended 1 or 2 sessions) | 31 (Attended 1 or 2 sessions)
Completed Intervention | 104 (Attended 3 or more sessions) | 104 (Attended 3 or more sessions)
Completed | 139 (Attended 3 or more sessions) | 135 (Attended 3 or more sessions)
Not Completed | 39 | 43
Not completed — 0 Sessions Attended | 34 | 37
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care | Total
Number analyzed (Participants) | 178 | 178 | 356
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 356 were randomized and analyzed.
  years | 34.7 (12.2) | 35 (11.3) | 34.9 (11.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Male | 146 | 153 | 299
  Gender Identity: Trans male/Trans man | 26 | 18 | 44
  Gender Identity: Other | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 17 | 16 | 33
  White | 129 | 134 | 263
  More than one race | 12 | 12 | 24
  Unknown or Not Reported | 0 | 2 | 2
Mental Health Treatment History [Count of Participants; unit: Participants]
  Treatment naive | 21 | 19 | 40
  Not treatment naive | 157 | 159 | 316
Depression (CES-D) [Mean (Standard Deviation); unit: units on a scale] — This is a 20-item questionnaire that asks about experience and frequency of depressive symptoms over the past week. Possible range of scores is 0-60, with the higher scores indicating the presence of more symptomatology. A score of 16 or higher identifies those individuals who are at risk for major depression (which is equivalent to endorsing at least 6 out of 20 symptoms for depression. Researchers will be looking for scores to reduce to below 16, indicating a lack of criteria being met for major depressive disorder.
  Baseline CESDs values reported, unadjusted for covariates.
  units on a scale | 30.61 (10.85) | 31.24 (10.81) | 30.92 (10.82)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Engage in Mental Health Treatment
Description: The number of participants who initiated mental health treatment/reinitiated mental health treatment versus those who did not. Mental health treatment engagement will be operationally defined as having ≥1 visit(s) or scheduled appointments to any mental health services within 120 days of the last online group.
Time Frame: Post-intervention (immediately following last online group), 60-day follow-up, and 120-day follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
Participants
  Post-Intervention | 23 | 18
  60-day follow-up | 31 | 26
  120-day follow-up | 28 | 31

2. Primary Outcome: Center for Epidemiological Studies Depression Scale
Description: This is a 20-item questionnaire that asks about experience and frequency of depressive symptoms over the past week. Possible range of scores is 0-60, with the higher scores indicating the presence of more symptomatology. A score of 16 or higher identifies those individuals who are at risk for major depression (which is equivalent to endorsing at least 6 out of 20 symptoms for depression. Researchers will be looking for scores to reduce to below 16, indicating a lack of criteria being met for major depressive disorder.
Time Frame: Baseline (pre-intervention), Post-intervention (immediately following last online group), 60-day follow-up, and 120-day follow-up.
Population: For outcome analyses, linear mixed models (LMM) of mental health symptoms were modeled as a repeated measures outcome variable, nested within participants, and nested within cohorts. Baseline values of the dependent variable, along with any baseline characteristics that differentiated the two groups, were included as time-invariant covariates (between participants), as was treatment group.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
score on a scale
  Baseline | 30.50 (.67) | 30.70 (.67)
  Post-intervention | 24.04 (.75) | 22.87 (.73)
  60-day follow-up | 27.33 (.77) | 25.46 (.75)
  120-day follow-up | 24.01 (.79) | 23.74 (.77)

3. Secondary Outcome: Post Traumatic Stress Disorder
Description: PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) , DSM-5 (PCL-5; Weathers et al., 2013) is a 20-item instrument that corresponds to the current psychiatric diagnostic criteria for PTSD. Participants respond on a Likert scale ranging from 0 (not at all) to 4 (extremely). A provisional PTSD diagnosis can be made by treating each item rated as 2 (moderately) or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 Criterion B item (Intrusion symptoms; questions 1-5), 1 Criterion C item (Avoidance symptoms; questions 6-7), 2 Criterion D items (Alternations in cognitions and mood; questions 8-14), 2 Criterion E items (Alterations in arousal and reactivity; questions 15-20). A PCL-5 cut-point of 33 appears to be a reasonable value to use for provisional PTSD diagnosis. Severity can be determined adding scores of each item together to determine a total score. The range is 0-80.
Time Frame: Baseline (immediately pre-intervention), Post-intervention (immediately following last online group), 60-day follow-up, and 120-day follow-up.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
score on a scale
  Baseline | 36.26 (.97) | 36.45 (.97)
  Post-intervention | 29.30 (1.10) | 27.84 (1.06)
  60-day follow-up | 32.22 (1.12) | 29.21 (1.10)
  120-day follow-up | 27.47 (1.14) | 25.57 (1.12)

4. Secondary Outcome: Psychosocial Functioning
Description: Inventory of Psychosocial Functioning (IPF-B; Rodriguez, Holowka, & Marx, 2012) is a brief 7-item scale that assesses functional impairment or quality of life related to trauma and PTSD. Questions assess for impairment in romantic relationships, family relationships, work, friendships and socializing, parenting, academic pursuits, and self-care. Higher scores indicate greater functional impairment. Respondents answer each item by using a 7-point scale ranging from 1 ("never") to 7 ("always"). The IPF yields an overall functional impairment score.
Time Frame: Baseline (immediately pre-intervention), Post-intervention (immediately following last online group), 60-day follow-up, and 120-day
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
score on a scale
  Baseline | 45.64 (1.36) | 44.71 (1.37)
  Post-intervention | 39.88 (1.56) | 38.51 (1.52)
  60-day follow-up | 39.97 (1.58) | 34.05 (1.56)
  120-day follow-up | 39.69 (1.62) | 38.72 (1.60)

5. Secondary Outcome: Substance Abuse
Description: The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) is an 8-item measure of use of alcohol, tobacco products, and other drugs across the lifespan and in the past 3 months. The test has been shown to be a valid indicator of active substance use with adequate construct validity. Scores are summed across for each drug category separately with a maximum score for tobacco = 31 and a maximum score for each of the other drug categories = 39. A Global Continuum of Risk Score can also be calculated by summing all items for all drug classes together with a maximum score of 414. Scores are categorized into Low (0 - 3), Moderate (4 - 26), and High (27+) risk.
Time Frame: Baseline (immediately pre-intervention)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
score on a scale
  Tobacco | 5.77 (.28) | 5.83 (.28)
  Alcohol | 8.83 (.35) | 8.93 (.35)
  Marijuana | 6.44 (.33) | 6.53 (.33)
  Cocaine | 1.58 (.17) | 1.69 (.17)
  Amphetamine/ Stimulant | 2.51 (.23) | 2.55 (.23)
  Inhalants | .96 (.15) | 1.06 (.15)
  Sedatives | 2.00 (.23) | 1.84 (.23)
  Hallucinogens | .98 (.15) | .98 (.15)
  Opioids | 1.02 (.17) | 1.03 (.17)
  Other | 8.83 (.35) | 8.93 (.35)
  Medical Marijuana | 1.68 (.30) | 1.65 (.30)

6. Secondary Outcome: Substance Abuse
Description: as for outcome 5
Time Frame: Post-intervention (immediately following last online group)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
Number analyzed (Participants) | 178 | 178
score on a scale
  Tobacco | 4.92 (.32) | 4.75 (.31)
  Alcohol | 7.71 (.40) | 8.26 (.39)
  Marijuana | 5.89 (.38) | 5.69 (.36)
  Cocaine | 1.39 (.20) | 1.04 (.19)
  Amphetamine/ Stimulant | 2.16 (.26) | 2.11 (.27)
  Inhalants | 1.06 (.16) | .90 (.17)
  Sedatives | 1.67 (.26) | 2.21 (.25)
  Hallucinogens | .88 (.17) | .98 (.17)
  Opioids | .83 (.19) | .99 (.19)
  Other | 4.92 (.32) | 4.75 (.31)
  Medical Marijuana | 1.55 (.39) | 2.74 (.36)

ADVERSE EVENTS:
Time Frame: From baseline to 120-day follow-up, approximately 170 days.
Arm/Group | Motivational Interviewing | MI With Trauma-informed SGM Affirmative Care
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/178
Serious Adverse Events (participants affected / at risk) | 2/178 | 0/178
Other Adverse Events (participants affected / at risk) | 5/178 | 12/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing (N=178) | MI With Trauma-informed SGM Affirmative Care (N=178)
Psychiatric hospitalization (Psychiatric disorders) | 1 (1) | 0 (0)
Sexual Assault (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing (N=178) | MI With Trauma-informed SGM Affirmative Care (N=178)
High Suicidality (Psychiatric disorders) | 5 (5) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT03794986/Prot_SAP_ICF_000.pdf